CLINICAL TRIAL: NCT01120860
Title: MRI and Decline of Aging Aviator Performance
Brief Title: Magnetic Resonance Imaging (MRI) and Decline of Aging Aviator Performance
Status: Completed | Type: Observational
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Joy Taylor, Clinical Professor (affiliated), Psychiatry & Behavioral Sciences, Stanford University
Other Study IDs: TAYRNW0001/TAY0002; 11097
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Age-related Cognitive Decline
Keywords: Cognitive Aging; Apolipoproteins E; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen genomic DNA
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MRI — MRI - routine imaging sequences, designed for anatomical quantification

SUMMARY:
The primary purpose of this study is to apply state-of-the-art Magnetic Resonance Imaging (MRI) and Magnetic Resonance Spectroscopic Imaging (MRSI) techniques to measure changes over time in the brain.

DETAILED DESCRIPTION:
We expect that MRI and MRSI techniques will be a useful adjunct in research efforts to understand individual differences in performance of a complex attention-demanding task, such as flying a plane or driving a car. Other predictors of change in performance of a complex task may include simple tests of processing speed and working memory, past training and recent practice of the task, and genetic risk factors for degenerative brain disease. In this project, we will examine whether baseline MR measures are as useful as longitudinal MR measures in predicting amount of change over time in task performance.

This research is part of a long-term effort to achieve earlier identification of individuals at risk of decline and ultimately minimize loss of function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included if they have participated in the protocol "Age-Related Longitudinal Changes in Aviator Performance" and agree to participate in this protocol.

Exclusion Criteria:

* Subjects will be excluded if they currently have a major neurological disease, unstable/untreated medical disease (such as untreated hypertension).
* In consideration of the magnetic fields in which subjects will be placed for the MR scanning, we will also exclude subjects who are unable to safely and comfortably complete the scanning session. This includes individuals who are wearing any metal prosthesis or who have cardiac pacemakers or any other nonremovable metal objects.
* Subjects reporting a history of severe claustrophobia or poorly controlled back pain will be excluded because it is unlikely they could comfortably remain still in the MRI scanner for the duration of the scan.
* In addition, subjects who do not fit in the apparatus will also be excluded.

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: active healthy pilots
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2002-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
flight simulator performance summary score | yearly for up to 6 years
  z-score composite of executing ATC communications, avoiding traffic, monitoring engine malfunctions, visual approach and landing

SECONDARY OUTCOMES:
CogScreen-AE | yearly
  computerized battery (assesses processing speed, executive function, paired assoc memory, n-back task, psychomotor tracking
Salthouse processing speed measures | yearl
  digit copy & pattern comparison

CONTACTS AND LOCATIONS:
Overall Officials: Joy Taylor, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States